CLINICAL TRIAL: NCT00199485
Title: Angelica Sinensis for the Treatment of Hot Flashes in Men Undergoing Androgen Deprivation Therapy for Prostate Cancer
Brief Title: Angelica Sinensis for the Treatment of Hot Flashes in Men Undergoing LHRH Therapy for Prostate Cancer
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's (Other)
Collaborators: St. Joseph's Health Care London (Other)
Responsible Party: Dr. Hassan Razvi, Lawson Health Research Institute
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: S-01-007; 08217
Record Dates: First submitted 2005-09-13; First posted 2005-09-20 (Estimated); Last update posted 2008-07-29 (Estimated); Status verified 2008-07

CONDITIONS: Prostate Cancer
Keywords: prostate cancer; Luteinizing Hormone Releasing Hormone; LHRH
MeSH Terms: conditions — Prostatic Neoplasms | interventions — angelicae sinensis extract

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): Angelica Sinensis
  Interventions: Drug: Angelica Sinensis
- 2 (Placebo Comparator): placebo
  Interventions: Drug: Angelica Sinensis

INTERVENTIONS:
Drug: Angelica Sinensis — Angelica Sinensis / placebo

SUMMARY:
Men undergoing androgen deprivation therapy for prostate cancer may experience significant side effects including symptoms of intense heat, facial flushing, and sweating. These so-called hot flashes are similar to those experienced by women during menopause. A traditional Chinese herbal preparation, Dong Quai, has been used for thousands of years to reduce the incidence and severity of hot flashes. Anecdotal evidence exists to support the use of Dong Quai in men treated with androgen deprivation therapy for prostate cancer.

Recently, the awareness and use of herbal remedies and over-the-counter preparations for a number of different conditions have increased dramatically. This trial was, therefore, designed to determine if Dong Quai significantly reduces the incidence and severity of hot flashes in men following androgen deprivation therapy for prostate cancer.

ELIGIBILITY:
Inclusion Criteria:

* Prostate cancer treated with some form of androgen deprivation therapy for at least one month. This includes either surgical (bilateral orchidectomy) or medical (LHRH agonist, pure or steroidal antiandrogen or combined) castration;
* Greater than seven vasomotor episodes per week;
* Significantly bothersome symptoms associated with these vasomotor episodes, which produce a desire in the patient to seek treatment to reduce both their incidence and severity;
* Documented informed consent to participate in the trial.

Exclusion Criteria:

* Enrolment in any other clinical trial or study protocol;
* Presence of pain due to prostate cancer;
* Life expectancy less than three months;
* Any severe concomitant condition that would make it undesirable, in the clinician's opinion, or the subject to participate in the trial or would jeopardize compliance with the trial protocol;
* Concomitant anticoagulation therapy or history of bleeding disorder or blood dyscrasia;
* Known hypersensitivity to Dong Quai.

Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 44 (Estimated)
Dates: Start 2002-10; Primary Completion 2008-06 (Actual); Study Completion 2008-06 (Actual)

PRIMARY OUTCOMES:
assess bone loss in men with prostate cancer being treated with LHRH | at each of 3 follow up visits

CONTACTS AND LOCATIONS:
Overall Officials: Hassan Razvi, MD, FRCSC, Principal Investigator — Urology, St. Joseph's Hospital, University of Western Ontario
Locations (1):
- Urology Clinic & Prostate Centre, St. Joseph's Hospital, St. Joseph's Health Care London, London, Ontario, Canada